CLINICAL TRIAL: NCT00002331
Title: A Randomized Open-Label Study of the Tolerability and Efficacy of Clarithromycin and Ethambutol in Combination With or Without Clofazimine for the Treatment of Disseminated MAC (dMAC) in Patients With AIDS
Brief Title: The Safety and Effectiveness of Clarithromycin Plus Ethambutol Used With or Without Clofazimine in the Treatment of MAC in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott (Industry)
Purpose: Treatment
Other Study IDs: 214A; M93-069
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2009-02

CONDITIONS: Mycobacterium Avium-intracellular Infection; HIV Infections
Keywords: Mycobacterium avium-intracellular Infection; Drug Therapy, Combination; Ethambutol; Clofazimine; Acquired Immunodeficiency Syndrome; Clarithromycin
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Ethambutol; Clarithromycin; Clofazimine

INTERVENTIONS:
Drug: Ethambutol hydrochloride
Drug: Clarithromycin
Drug: Clofazimine

SUMMARY:
PRIMARY: To assess the tolerability of the combination regimen of clarithromycin plus ethambutol with or without clofazimine in patients with disseminated Mycobacterium avium Complex (dMAC).

SECONDARY: To determine the proportion of patients achieving a sterile blood culture along with the time required to achieve it. To determine the duration of bacteriological response, defined as length of time that blood cultures remain sterile.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* History of HIV seropositivity.
* Disseminated MAC.
* Positive blood culture for MAC within 4 weeks prior to study entry.
* Consent of parent or guardian if less than 18 years of age.
* Ability to complete the study.

NOTE:

* Patients with active opportunistic infections other than dMAC are permitted if dosage and clinical parameters have been stable for 4 weeks prior to enrollment.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Active therapy with carbamazepine or theophylline, unless investigator agrees to carefully monitor blood levels.
* Active therapy with investigational drugs other than treatment for HIV disease, except with approval of the sponsor.
* Concomitant terfenadine (Seldane or Seldane-D) or astemizole (Hismanal).
* Amikacin.
* Azithromycin.
* Capreomycin.
* Ciprofloxacin.
* Cycloserine.
* Ethionamide.
* Gentamicin.
* Kanamycin.
* Levofloxacin.
* Lomefloxacin.
* Ofloxacin.
* Rifampin.
* Rifabutin.
* Sparfloxacin.
* Streptomycin.
* Any other aminoglycosides, quinolones, and macrolides.

Patients with the following prior conditions are excluded:

History of allergy or hypersensitivity to macrolides, ethambutol, or clofazimine.

Prior Medication:

Excluded:

* Other antimycobacterials, including aminoglycosides, ansamycin (rifabutin), other macrolides (such as clindamycin), quinolones, and rifampin, between screening and study entry.
* Clarithromycin or azithromycin as prophylaxis or treatment (for any cause) for more than 14 days cumulative within the past 2 months.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-01; Primary Completion 1995-03 (Actual); Study Completion 1995-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (17):
  - Kaiser Permanente Med Ctr, Los Angeles, California
  - UCD Med Ctr, Sacramento, California
  - Kaiser Permanente Med Ctr, San Francisco, California
  - Santa Clara Valley Med Ctr, San Jose, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Dr Margaret Fischel, Miami, Florida
  - Saint Joseph's Hosp / Infectious Disease Rsch Institute, Tampa, Florida
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Tulane Univ Med School, New Orleans, Louisiana
  - Johns Hopkins Univ School of Medicine, Baltimore, Maryland
  - Beth Israel Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Dr Stephen Hauptman, Philadelphia, Pennsylvania
  - Vanderbilt Univ School of Medicine, Nashville, Tennessee
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Houston Veterans Administration Med Ctr, Houston, Texas
- Dr Javier Morales, Condado San Juan, Puerto Rico

REFERENCES:
- [Background] Chaisson RE, Keiser P, Pierce M, Fessel WJ, Ruskin J, Lahart C, Benson CA, Meek K, Siepman N, Craft JC. Clarithromycin and ethambutol with or without clofazimine for the treatment of bacteremic Mycobacterium avium complex disease in patients with HIV infection. AIDS. 1997 Mar;11(3):311-7. doi: 10.1097/00002030-199703110-00008. PMID 9147422